CLINICAL TRIAL: NCT04973670
Title: Protective Effect of Sivelestat Sodium on ARDS in Patients With Sepsis: Multicenter, Random, Double-blind, Parallel, Placebo Control Clinical Trials
Brief Title: Protective Effect of Sivelestat Sodium on ARDS in Patients With Sepsis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Ling Liu, professor, Southeast University, China
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ZDHL
Record Dates: First submitted 2021-07-13; First posted 2021-07-22 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-04

CONDITIONS: ARDS
Keywords: Sepsis; Respiratory Failure; ARDS; efficacy; Sivelestat sodium
MeSH Terms: conditions — Sepsis; Respiratory Insufficiency

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sivelestat sodium (Experimental): Sivelestat sodium 0.2mg/kg.h
  Interventions: Drug: Sivelestat sodium
- placebo (Active Comparator): The same amount of NS containing only sivelestat sodium excipients
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sivelestat sodium — Sivelestat sodium 0.2mg/kg.h for 1-7 days
  Arms: Sivelestat sodium
Drug: Placebo — The same amount of NS containing only sivelestat sodium excipients
  Arms: placebo

SUMMARY:
Sivelestat sodium has been approved for use in patients with SIRS and ALI, but whether it can protect patients with sepsis from developing ARDS remains unknown.The aim of this study was to determine whether sivelestat sodium has a protective effect on ARDS in patients with sepsis.

DETAILED DESCRIPTION:
The study was conducted in accordance with good clinical practice and with the guidelines set out in the Declaration of Helsinki. After approval from local and national ethics committees, patients from 3 centers in China were recruited.

All patients were randomized, in a double-blind manner, to receive either sivelestat sodium regimen or a placebo regimen for 1- 7 days in ICU.

The aim of this study was to determine whether sivelestat sodium has a protective effect on ARDS in patients with sepsis.

ELIGIBILITY:
Inclusion Criteria:

* Within 24 hours after admission, sepsis 3.0 diagnostic criteria were met;
* The patients or their family members fully understand the purpose and significance of the trial, voluntarily participate in the clinical trial, and sign the informed consent.

Exclusion Criteria:

* Patients with ARDS were identified at the time of admission;
* Patients who explicitly refused mechanical ventilation;
* Patients with 3 or more extrapulmonary organ injuries and organ failure(single organ SOFA score ≥ 3);
* Patients who need home oxygen therapy or with home mechanical ventilation (by tracheotomy or noninvasive ventilation, but excluding CPAP / BiPAP, only for patients with obstructive sleep apnea);
* The patient whose expected survival time was less than 48 hours;
* Pregnant women and lactating women;
* Other conditions judged by the researcher not suitable for inclusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Estimated)
Dates: Start 2021-10-11 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
Progression to ARDS within 7 days (Berlin criteria) | From study drug administration to days 7
  The proportion of patients with sepsis progressing to ARDS

SECONDARY OUTCOMES:
Oxygenation index (PaO2/FiO2) or SpO2 / FiO2 on day 1, 3 and 7 from drug administration | From study drug administration to days 7
  PaO2/FiO2 or SpO2 / FiO2 was recorded on day 1, 3 and 7 from drug administration
Concentration of inflammatory factors on day 1, 3 and 7 from drug administration | From study drug administration to days 7
  Inflammatory factors include Interleukin(IL)-1β,IL-6, IL-8, IL-10, tumor necrosis factor(TNF)-α
Concentration of neutrophil elastase on day 1, 3 and 7 from drug administration | From study drug administration to days 7
  Concentration of neutrophil elastase was recorded on day 1, 3 and 7 from drug administration
Platelet count on day 1, 3 and 7 from drug administration | From study drug administration to days 7
  Platelet count was recorded on day 1, 3 and 7 from drug administration
Concentration of C-reactive protein on day 1, 3 and 7 from drug administration | From study drug administration to days 7
  Concentration of High sensitivity C-reactive protein was recorded on day 1, 3 and 7 from drug administration
Sequential organ failure assessment (SOFA) score on day 1, 3 and 7 from drug administration | From study drug administration to days 7
  The SOFA scores on day 1, 3 and 7 were recorded
The 28-day ventilator-free days (VFD) | From study drug administration to day 28
  Days alive and free from mechanical ventilation from study drug administration to day 28
The 28-day shock-free days | From study drug administration to day 28
  Days alive and free from vasopressor support which define as infusion of any vasopressor/inotrope agent for a minimum of 1 hour (i.e.norepinephrine, epinephrine, phenylephrine, vasopressin analogues, angiotensin, dopamine, dobutamine, milrinone or levosimendan) from study drug administration to day 28
The 28-day time to clinical improvement | From study drug administration to day 28
  Defined as the time from randomization to an improvement of two points (from the status at randomization) on a seven-category ordinal scale or live discharge from the hospital, whichever came first. The seven-category ordinal scale consisted of the following categories: 1, not hospitalized with resumption of normal activities; 2, not hospitalized, but unable to resume normal activities; 3, hospitalized, not requiring supplemental oxygen; 4, hospitalized, requiring supplemental oxygen; 5, hospitalized, requiring nasal high-flow oxygen therapy, noninvasive mechanical ventilation, or both; 6, hospitalized, requiring ECMO, invasive mechanical ventilation, or both; and 7, death.
Length of hospital stay | From administration to discharge hospital, up to 90 days
  The number of days the subject stayed in the hospital
The 28-day mortality | From study drug administration to day 28
  Death of any cause from study drug administration to day 28
The 90-day mortality | From study drug administration to day 90
  Death of any cause from study drug administration to day 90

CONTACTS AND LOCATIONS:
Overall Officials: Liu ling, MD, Study Chair — Department of Critical Care Medicine, Zhongda Hospital, School of Medicine, Southeast University
Locations (1):
- Nanjing Zhong-Da Hospital, Southeast University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ma S, Li C, Gao Z, Xie J, Qiu H, Yang Y, Liu L. Effects of intravenous sivelestat sodium on prevention of acute respiratory distress syndrome in patients with sepsis: study protocol for a double-blind multicentre randomised controlled trial. BMJ Open. 2023 Sep 13;13(9):e074756. doi: 10.1136/bmjopen-2023-074756. PMID 37709320